CLINICAL TRIAL: NCT04985344
Title: Treatment of Pediatric Post-traumatic Stress Disorder With Memory Reactivation Under the Influence of Propranolol: A Randomized Placebo-controlled Trial. PPP
Brief Title: Treatment of Pediatric Post-traumatic Stress Disorder With Memory Reactivation Under the Influence of Propranolol
Acronym: PPP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/18/0471; 2020-005956-39 (EudraCT Number)
Record Dates: First submitted 2021-07-21; First posted 2021-08-02 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: PTSD
Keywords: PTSD; traumatic memory reactivation; pediatric; Propranolol; Post-traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propranolol (Experimental): Patient will receive oral propranolol
  Interventions: Drug: Propranolol Oral Product; Other: memory reactivation
- Placebo (Placebo Comparator): Patient will receive oral placebo
  Interventions: Drug: Placebo; Other: memory reactivation

INTERVENTIONS:
Drug: Propranolol Oral Product — Child will receive oral propranolol (syrup). The dose of propranolol will increase gradually over the first 3 treatment sessions in order to assess tolerance.
  Other Names: Propranolol
  Arms: Propranolol
Drug: Placebo — Child will receive oral placebo (syrup). The dose of placebo will increase gradually over the first 3 treatment sessions in order to match propranolol intervention.
  Arms: Placebo
Other: memory reactivation — 90 minutes after the propranolol take, a trained psychologist will ask the child to recount his trauma.

SUMMARY:
By age 18, roughly 8% of traumatized youth have met criteria for a diagnosis of PTSD, with numbers rising up to 40% in cases of sexual abuse and assault. To date there is no empirical support for the use of psychopharmacological interventions as treatment of pediatric PTSD. Trauma-focused psychotherapeutic/TFP approaches should be favored in childhood PTSD. However, when compared to active control conditions, TFP produced a mean effect size on child and adolescents population (g=0.83). Moreover, in therapies with a substantial exposure component, the intense and lengthy reexperiencing of the traumatic event results in a substantial proportion of participants dropping out.

The reactivation of a previously consolidated memory can make it labile, subsequently requiring a re-stabilization of it called reconsolidation of the memory.

Acting on these reconsolidation processes makes possible to interfere with the subsequent storage of this memory.

DETAILED DESCRIPTION:
By age 18, roughly 8% of traumatized youth have met criteria for a diagnosis of PTSD, with numbers rising up to 40% in cases of sexual abuse and assault. To date there is no empirical support for the use of psychopharmacological interventions as treatment of pediatric PTSD. Trauma-focused psychotherapeutic/TFP approaches should be favored in childhood PTSD. However, when compared to active control conditions, TFP produced a mean effect size on child and adolescents population (g=0.83). Moreover, in therapies with a substantial exposure component, the intense and lengthy reexperiencing of the traumatic event results in a substantial proportion of participants dropping out.

The reactivation of a previously consolidated memory can make it labile, subsequently requiring a re-stabilization of it called reconsolidation of the memory.

Acting on these reconsolidation processes makes possible to interfere with the subsequent storage of this memory.

The combination of the targeted reactivation of the traumatic memory and the intake of an agent that decreases the reconsolidation can thus disrupt the recall of unwanted memories and thus serve as a treatment for people suffering from traumatic memories, such as in PTSD.

Since stimulation of β-noradrenergic receptors facilitates the consolidation of memories as well as their re-consolidation, an antagonist of these receptors, propranolol, has generated considerable interest as a treatment to alleviate emotional and traumatic memories in individuals with PTSD.

In adults diagnosed with long-standing PTSD two 6-week, double-blind, placebocontrolled, randomised clinical trials, one in 60 subjects and the other in 67 have shown promising results. PTSD participants who actively recalled their traumatic event under the influence of propranolol once a week for up to 6 weeks showed a substantial decrease in symptom ratings compared with placebo. Thus, all of this data led the team to propose a comparable design study in children with PTSD

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-12 years
* CPTS-RI total score ≥40
* Primary diagnosis of PTSD (6 months or more after the traumatic event)
* Heart rate ≥ 55 bpm
* Systolic blood pressure ≥ 95 mm Hg
* Affiliation to a social security scheme
* Written consent signed by the parents/holders of parental authority and the investigator
* Acceptance of the protocol by the child-Child and Parents/Holders of parental authority fluent in French

Exclusion Criteria:

* Age<7 years or ≥13 years
* Children whose parents have been deprived of their authority
* Contraindication to propranolol (cardiogenic shock, sinus bradycardia, hypotension (< fifth percentile oscillometric or <2SD) (Banker et al., 2016 - see APPENDIX 1), greater than first-degree heart block, heart failure, bronchial asthma and hypersensitivity to propranolol hydrochloride)
* Concurrent medication with possible interactions with propranolol (cf 8.2)
* Concurrent psychotropic drugs that have been shown to be effective in improving symptoms of PTSD (Antidepressants, atypical antipsychotics, mood stabilizers)
* Concurrent psychotherapy (>1 structured session/month declared by the clinician who follows the child)
* Current active psychosis, anorexia nervosa, bulimia nervosa, binge-eating disorder, attention-deficit hyperactivity disorder, autism spectrum disorder
* Children with psoriasis
* Children with a predisposition to hypoglycemia
* Obsessive-compulsive disorders
* Bipolar Disorders
* Mental retardation,
* Traumatic brain injury (loss of consciousness > 10 minutes)
* Currently treated with a bradycardic drug
* Concurrent participation to another interventional study
* Renal or Hepatic Impairment
* Pregnancy

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Child Post-Traumatic Stress Reaction Index/CPTS-RI | week 8
  The main evaluation criterion will be the difference between the Child Post-Traumatic Stress Reaction Index/CPTS-RI total score administered at week 8 and week 0. The CPTS-RI is a scale comprised of 20 Likert-type items, intended for children from 6 to 16 years, which evaluates the symptoms of PTSD after exposure to various traumatic events. Each item frequency is rated on a 5-point scale, from never (=0) to almost always (=4). The global score consists of the sum of the 20 items and ranges from 0 to 80, with higher scores indicating higher PTSD symptom severity. The time required for completion of the scale is 15-20 min. A total score of 12-24 is associated with a mild level of PTSD, from 25-39 with a moderate level, from 40-59 with a severe level, and ≥60 with a very severe level.

SECONDARY OUTCOMES:
Child Post-Traumatic Stress Reaction - Week 32 Index/CPTS-RI | week 32
  The difference between the Child Post-Traumatic Stress Reaction Index/CPTS-RI total score at week 32 and week 8 . The CPTS-RI is a scale comprised of 20 Likert-type items, intended for children from 6 to 16 years, which evaluates the symptoms of PTSD after exposure to various traumatic events. Each item frequency is rated on a 5-point scale, from never (=0) to almost always (=4). The global score consists of the sum of the 20 items and ranges from 0 to 80, with higher scores indicating higher PTSD symptom severity. The time required for completion of the scale is 15-20 min. A total score of 12-24 is associated with a mild level of PTSD, from 25-39 with a moderate level, from 40-59 with a severe level, and ≥60 with a very severe level.
Child Post-Traumatic Stress Reaction - Week 60 Index/CPTS-RI | week 60
  The difference between the Child Post-Traumatic Stress Reaction Index/CPTS-RI total score administered at week 60 and week 8. The CPTS-RI is a scale comprised of 20 Likert-type items, intended for children from 6 to 16 years, which evaluates the symptoms of PTSD after exposure to various traumatic events. Each item frequency is rated on a 5-point scale, from never (=0) to almost always (=4). The global score consists of the sum of the 20 items and ranges from 0 to 80, with higher scores indicating higher PTSD symptom severity. The time required for completion of the scale is 15-20 min. A total score of 12-24 is associated with a mild level of PTSD, from 25-39 with a moderate level, from 40-59 with a severe level, and ≥60 with a very severe level.
Child PTSD Checklist-Child version/CPC-C total score | Week 8
  The difference between the Child PTSD Checklist-Child version/CPC-C total score administered at week 8 and week 0 on items 14-34. The CPC-C includes a traumatic events page, 21 PTSD symptoms and 6 items of functional impairment. It is free in the public domain. For scoring the CPC-C 7-18 years (Version May 23, 2014.), the Traumatic Events page (items 1-13) is important to include before administering the symptom portion. Items 14-34 are PTSD symptom items.
Child PTSD Checklist-Child version/CPC-C total score - Week 32 | Week 32
  The difference between the Child PTSD Checklist-Child version/CPC-C total score administered at week 8 and week 32 on items 14-34. The CPC-C includes a traumatic events page, 21 PTSD symptoms and 6 items of functional impairment. It is free in the public domain. For scoring the CPC-C 7-18 years (Version May 23, 2014.), the Traumatic Events page (items 1-13) is important to include before administering the symptom portion. Items 14-34 are PTSD symptom items.
Child PTSD Checklist-Child version/CPC-C total score - Week 60 | Week 60
  The difference between the Child PTSD Checklist-Child version/CPC-C total score administered at week 8 and week 60 on items 14-34. The CPC-C includes a traumatic events page, 21 PTSD symptoms and 6 items of functional impairment. It is free in the public domain. For scoring the CPC-C 7-18 years (Version May 23, 2014.), the Traumatic Events page (items 1-13) is important to include before administering the symptom portion. Items 14-34 are PTSD symptom items.
Child PTSD Checklist-Parent version/CPC-P total score - Week 32 | Week 32
  The difference between the Child PTSD Checklist-Parent version/CPC-P total score administered at week 8 and week 32 on items 14-34 (PTSD symptom items). The CPC-P includes a traumatic events page, 21 PTSD symptoms and 6 items of functional impairment. It is free in the public domain. For scoring the CPC-P, 7-18 years (Version May 23, 2014.), the Traumatic Events page (items 1-13) is important to include before administering the symptom portion. Items 14-34 are PTSD symptom items.
Child PTSD Checklist-Parent version/CPC-P total score - Week 60 | Week 60
  The difference between the Child PTSD Checklist-Parent version/CPC-P total score administered at week 8 and week 60 on items 14-34 (PTSD symptom items). The CPC-P includes a traumatic events page, 21 PTSD symptoms and 6 items of functional impairment. It is free in the public domain. For scoring the CPC-P, 7-18 years (Version May 23, 2014.), the Traumatic Events page (items 1-13) is important to include before administering the symptom portion. Items 14-34 are PTSD symptom items.
Child PTSD Checklist-Parent version/CPC-P total score | Week 8
  The difference between the Child PTSD Checklist-Parent version/CPC-P total score administered at week 8 and week 0 on items 14-34 (PTSD symptom items). The CPC-P includes a traumatic events page, 21 PTSD symptoms and 6 items of functional impairment. It is free in the public domain. For scoring the CPC-P, 7-18 years (Version May 23, 2014.), the Traumatic Events page (items 1-13) is important to include before administering the symptom portion. Items 14-34 are PTSD symptom items.
Kiddie-SADS-Present and Lifetime Version DSM-5/K-SADS-PL-DSM5 | week 8
  The percentage of children without a current diagnosis of PTSD assessing with Kiddie-SADS-Present and Lifetime Version DSM-5/K-SADS-PL-DSM5. The K-SADS-PL-DSM5 (November 2016) is a semi-structured diagnostic interview designed to collect information from the child or adolescent as well as their parents or other informants.
Current diagnosis of PTSD at Week 32 | week 32
  The percentage of children without a current diagnosis of PTSD assessing with Kiddie-SADS-Present and Lifetime Version DSM-5/K-SADS-PL-DSM5. The K-SADS-PL-DSM5 (November 2016) is a semi-structured diagnostic interview designed to collect information from the child or adolescent as well as their parents or other informants.
Children Depression Inventory/CDI total score | week 8
  The difference between the Children Depression Inventory/CDI total score administered at week 8 and week 0. The CDI is comprised of 27 items assessing self-reported symptoms of depression in children and adolescents 7-17 years of age.
Children Depression Inventory/CDI total score - Week 32 | week 32
  The difference between the Children Depression Inventory/CDI total score administered at week 8 and week 32. The CDI is comprised of 27 items assessing self-reported symptoms of depression in children and adolescents 7-17 years of age.
Children Depression Inventory/CDI total score - Week 60 | week 60
  The difference between the Children Depression Inventory/CDI total score administered at week 8 and week 60. The CDI is comprised of 27 items assessing self-reported symptoms of depression in children and adolescents 7-17 years of age.
Children's Sleep Habits Questionnaire/CSHQ Parent version total score | week 8
  The difference between the Children's Sleep Habits Questionnaire/CSHQ Parent version total score administered at week 8 and week 0.The CSHQ was designed by clinical researchers at Brown University for children aged 4 through 12 years, to screen for the most common sleep problems in that age group.The first column 'of responses are scored: Usually=3, Sometimes=2, Rarely=1 for the entire questionnaire (except for the R=reversed items, which are considered to be "desirable" sleep behaviors, and thus scored in the opposite direction)
Children's Sleep Habits Questionnaire/CSHQ Parent version total score - Week 32 | week 32
  The difference between the Children's Sleep Habits Questionnaire/CSHQ Parent version total score administered at week 8 and week 32.The CSHQ was designed by clinical researchers at Brown University for children aged 4 through 12 years, to screen for the most common sleep problems in that age group.The first column 'of responses are scored: Usually=3, Sometimes=2, Rarely=1 for the entire questionnaire (except for the R=reversed items, which are considered to be "desirable" sleep behaviors, and thus scored in the opposite direction)
Children's Sleep Habits Questionnaire/CSHQ Parent version total score - Week 60 | week 60
  The difference between the Children's Sleep Habits Questionnaire/CSHQ Parent version total score administered at week 8 and week 60.The CSHQ was designed by clinical researchers at Brown University for children aged 4 through 12 years, to screen for the most common sleep problems in that age group.The first column 'of responses are scored: Usually=3, Sometimes=2, Rarely=1 for the entire questionnaire (except for the R=reversed items, which are considered to be "desirable" sleep behaviors, and thus scored in the opposite direction)
Comorbidity of other mental disorders | week 8
  Using the K-SADS-PL DSM-5
Corsi Blocks task | week 8
  The difference between the Corsi blocks task administered at week 0 and at week 8. The Corsi Blocks task assesses the visuospatial component of working memory but uses various cognitive processes. The subject needs to reproduce, in the same or reverse order, a sequence of pointing movements to different cubes shown by the rater
CGAS Children's Global Assessment Scale total score | week 32
  The difference between the CGAS Children's Global Assessment Scale total score administered at week 8 and the score administered at week 32. The Childrens Global Assessment Scale (CGAS) is a measure developed by Schaffer and colleagues at the Department of Psychiatry, Columbia University to provide a global measure of level of functioning in children and adolescents. The measure provides a single global rating only, on scale of 0-100.
CGAS Children's Global Assessment Scale total score - Week 60 | week 60
  The difference between the CGAS Children's Global Assessment Scale total score administered at week 8 and the score administered at week 60. The Childrens Global Assessment Scale (CGAS) is a measure developed by Schaffer and colleagues at the Department of Psychiatry, Columbia University to provide a global measure of level of functioning in children and adolescents. The measure provides a single global rating only, on scale of 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Birmes, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olliac B, Birmes P, Bui E, Allenou C, Brunet A, Claudet I, Sales de Gauzy J, Grandjean H, Raynaud JP. Validation of the French version of the Child Post-Traumatic Stress Reaction Index: psychometric properties in French speaking school-aged children. PLoS One. 2014 Dec 2;9(12):e112603. doi: 10.1371/journal.pone.0112603. eCollection 2014. PMID 25460912
- [Background] Roullet P, Vaiva G, Very E, Bourcier A, Yrondi A, Dupuch L, Lamy P, Thalamas C, Jasse L, El Hage W, Birmes P. Traumatic memory reactivation with or without propranolol for PTSD and comorbid MD symptoms: a randomised clinical trial. Neuropsychopharmacology. 2021 Aug;46(9):1643-1649. doi: 10.1038/s41386-021-00984-w. Epub 2021 Feb 21. PMID 33612830
- [Background] Birmes P, Raynaud JP, Daubisse L, Brunet A, Arbus C, Klein R, Cailhol L, Allenou C, Hazane F, Grandjean H, Schmitt L. Children's enduring PTSD symptoms are related to their family's adaptability and cohesion. Community Ment Health J. 2009 Aug;45(4):290-9. doi: 10.1007/s10597-008-9166-3. Epub 2009 Jul 21. PMID 19621258